CLINICAL TRIAL: NCT01799889
Title: A Phase 2, Open-Label Study Evaluating the Efficacy, Safety, Tolerability, and Pharmacodynamics of GS-9973 in Subjects With Relapsed or Refractory Hematologic Malignancies
Brief Title: Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacodynamics of Entospletinib in Adults With Relapsed or Refractory Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision to discontinue development of entospletinib.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-339-0102
Record Dates: First submitted 2013-02-13; First posted 2013-02-27 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Chronic Lymphocytic Leukemia; Mantle Cell Lymphoma; Diffuse Large B-cell Lymphoma; Non-FL Indolent Non-Hodgkin's Lymphoma; Follicular Lymphoma
Keywords: SYK inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — 6-(1H-indazol-6-yl)-N-(4-morpholinophenyl)imidazo(1,2-a)pyrazin-8-amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- CLL, Entospletinib MM/SDD (Experimental): Participants with CLL, receive original formulation (mono-mesylate [MM]) of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib (spray dried dispersion [SDD]) 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib MM; Drug: Entospletinib SDD
- FL, Entospletinib MM/SDD (Experimental): Participants with FL, receive original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib MM; Drug: Entospletinib SDD
- DLBCL, Entospletinib MM/SDD (Experimental): Participants with DLBCL, receive original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib MM; Drug: Entospletinib SDD
- MCL, Entospletinib MM/SDD (Experimental): Participants with MCL, receive original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib MM; Drug: Entospletinib SDD
- non-FL iNHL, Entospletinib MM/SDD (Experimental): Participants with non-FL iNHL (ie, participants with LPL/WM, SLL, or MZL), receive original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib MM; Drug: Entospletinib SDD
- CLL; Prior BCR Inhibitor Naive, Entospletinib SDD 100 mg (Experimental): Participants with CLL, who are prior B-cell receptor (BCR) inhibitor naive, receive new formulation of entospletinib 100 mg (1 × 100 mg tablet) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD
- CLL; Prior BCR Inhibitor Naive, Entospletinib SDD 200 mg (Experimental): Participants with CLL, who are prior BCR inhibitor naive, receive new formulation of entospletinib 200 mg (1 × 200 mg tablet) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD
- CLL; Prior BCR Inhibitor Naive, Entospletinib SDD 400 mg (Experimental): Participants with CLL, who are prior BCR inhibitor naive, receive new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD
- CLL (Non-Richters) Prior BTK Inhibitor, Entospletinib SDD (Experimental): Participants with CLL and simple progression (non-Richters), who are exposed to Bruton tyrosine kinase (BTK) inhibitor, receive new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD
- CLL (Non-Richters) Prior PI3K Inhibitor, Entospletinib SDD (Experimental): Participants with CLL and simple progression (non-Richters), who are exposed to phosphatidylinositol 3-kinase (PI3K) inhibitor, receive new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD
- CLL (Richters) Prior BTK Inhibitor, Entospletinib SDD (Experimental): Participants with CLL, who transform to Richters or Richters-like syndrome and are exposed to BTK inhibitor, receive new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD
- CLL (Richters) Prior PI3K Inhibitor, Entospletinib SDD (Experimental): Participants with CLL, who transform to Richters or Richters-like syndrome and are exposed to PI3K inhibitor, receive new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib will continue until disease progression or unacceptable toxicity.
  Interventions: Drug: Entospletinib SDD

INTERVENTIONS:
Drug: Entospletinib MM — Entospletinib MM tablet administered orally
  Other Names: GS-9973
  Arms: CLL, Entospletinib MM/SDD; DLBCL, Entospletinib MM/SDD; FL, Entospletinib MM/SDD; MCL, Entospletinib MM/SDD; non-FL iNHL, Entospletinib MM/SDD
Drug: Entospletinib SDD — Entospletinib SDD tablet administered orally
  Other Names: GS-9973 SDD

SUMMARY:
The primary objective of the study is to evaluate efficacy of entospletinib in participants with relapsed or refractory hematologic malignancies. Participants with the following relapsed or refractory hematologic malignancies will be enrolled into the study: relapsed or refractory chronic lymphocytic leukemia (CLL), mantle cell lymphoma (MCL), diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), or non-FL indolent non-Hodgkin lymphomas (iNHL; including lymphoplasmacytoid lymphoma/ Waldenström macroglobulinemia [LPL/WM], small lymphocytic lymphoma [SLL], or marginal zone lymphoma [MZL]).

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of B-cell iNHL, DLBCL, MCL, or CLL as documented by medical records and with histology based on criteria established by the World Health Organization
* For institutions that have Phase 3 or Phase 4 protocols studying idelalisib (Zydelig®) ; individuals with malignancies being studied in these protocols must have failed screening in the respective idelalisib protocol
* Prior treatment for lymphoid malignancy requiring treatment for progressive disease
* Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy
* All acute toxic effects of any prior antitumor therapy resolved to Grade ≤ 1 before the start of study drug
* Karnofsky performance status of ≥ 60
* Life expectancy of at least 3 months

Key Exclusion Criteria:

* Known histological transformation from iNHL or CLL to an aggressive form of non-Hodgkin lymphoma (ie, Richter transformation) except if the CLL participant is enrolling in the BCR previously treated cohort
* Known active central nervous system or leptomeningeal lymphoma
* Presence of known intermediate- or high-grade myelodysplastic syndrome
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of start of study drug
* Ongoing liver injury
* Ongoing or recent hepatic encephalopathy
* Ongoing drug-induced pneumonitis
* Ongoing inflammatory bowel disease
* Ongoing alcohol or drug addiction
* Pregnancy or breastfeeding
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy
* Concurrent participation in an investigational drug trial with therapeutic intent

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (48):
- United States (46):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Oncology Associates, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Sharp Memorial Hospital, San Diego, California
  - Rocky Mountain Cancer Centers, LLP, Boulder, Colorado
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Florida Cancer - Colonial, Fort Myers, Florida
  - Memorial Cancer Institute, Hollywood, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Northside Hospital, Atlanta, Georgia
  - Gwinnett Hospital System Dba The Center for Cancer Care, Lawrenceville, Georgia
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Hematology Oncology Clinic, PLLC, Baton Rouge, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Oncology Hematology West PC dba Nebraska Cancer Specialists, Omaha, Nebraska
  - One Medical Center Drive, Lebanon, New Hampshire
  - Summit Medical Group, P.A., Florham Park, New Jersey
  - Clinical Research Alliance, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Williamette Valley Cancer Center and Research Institute, Springfield, Oregon
  - Prairie Lakes Health Care System, Inc., Watertown, South Dakota
  - Jones Clinic PC, Germantown, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Cancer Care Network of South Texas, San Antonio, Texas
  - Cancer Care Center of South Texas, San Antonio, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Columbia Basin Hematology and Oncology, Kennewick, Washington
  - University of Washington, Seattle, Washington
  - Northwest Cancer Specialists, PC, Vancouver, Washington
  - Yakima Valley Memorial Hospital North Star Lodge, Yakima, Washington
- Canada (2):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sir Mortimer B. Davis-Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharman J, Hawkins M, Kolibaba K, Boxer M, Klein L, Wu M, Hu J, Abella S, Yasenchak C. An open-label phase 2 trial of entospletinib (GS-9973), a selective spleen tyrosine kinase inhibitor, in chronic lymphocytic leukemia. Blood. 2015 Apr 9;125(15):2336-43. doi: 10.1182/blood-2014-08-595934. Epub 2015 Feb 18. PMID 25696919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States and Canada. The first participant was screened on 14 March 2013. The last study visit occurred on 30 January 2020.
Pre-assignment Details: 444 participants were screened.
Groups:
- CLL: Entospletinib MM/SDD: Participants with chronic lymphocytic leukemia (CLL), received original formulation (mono-mesylate [MM]) of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib (spray dried dispersion [SDD]) 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- FL: Entospletinib MM/SDD: Participants with follicular lymphoma (FL), received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- DLBCL: Entospletinib MM/SDD: Participants with diffuse large B-cell lymphoma (DLBCL), received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- MCL: Entospletinib MM/SDD: Participants with mantle cell lymphoma (MCL), received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- Non-FL iNHL: Entospletinib MM/SDD: Participants with non-FL indolent non-Hodgkin lymphomas (iNHL), (ie, participants with lymphoplasmacytoid lymphoma/ waldenström macroglobulinemia [LPL/WM], small lymphocytic lymphoma [SLL], or marginal zone lymphoma [MZL]), received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg: Participants with CLL, who were prior B-cell receptor (BCR) inhibitor naive, received new formulation of entospletinib 100 mg (1 × 100 mg tablet) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg: Participants with CLL, who were prior BCR inhibitor naive, received new formulation of entospletinib 200 mg (1 × 200 mg tablet) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg: Participants with CLL, who were prior BCR inhibitor naive, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD: Participants with CLL and simple progression (non-Richters), who were exposed to Bruton tyrosine kinase (BTK) inhibitor, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD: Participants with CLL and simple progression (non-Richters), who were exposed to phosphatidylinositol 3-kinase (PI3K) inhibitor, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD: Participants with CLL, who transformed to Richters or Richters-like syndrome and were exposed to BTK inhibitor, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD: Participants with CLL, who transformed to Richters or Richters-like syndrome and were exposed to PI3K inhibitor, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Started | 41 | 41 | 44 | 39 | 49 | 20 | 21 | 20 | 33 | 8 | 7 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 41 | 41 | 44 | 39 | 49 | 20 | 21 | 20 | 33 | 8 | 7 | 3
Not completed — Adverse Event | 4 | 4 | 5 | 1 | 11 | 1 | 5 | 2 | 3 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 5 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 4 | 4 | 5 | 5 | 5 | 2 | 6 | 0 | 0 | 1
Not completed — Progressive Disease | 30 | 26 | 25 | 30 | 23 | 9 | 8 | 13 | 18 | 5 | 3 | 1
Not completed — Specified Criteria for Withdrawal | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 6 | 4 | 0 | 5 | 1 | 3 | 1 | 2 | 1 | 1 | 1
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all enrolled participants who took at least one dose of study drug with treatment group designated according to the planned treatment.
Groups:
- CLL: Entospletinib MM/SDD: Participants with CLL, received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- FL: Entospletinib MM/SDD: Participants with FL, received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- DLBCL: Entospletinib MM/SDD: Participants with DLBCL, received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- MCL: Entospletinib MM/SDD: Participants with MCL, received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- Non-FL iNHL: Entospletinib MM/SDD: Participants with iNHL (ie, participants with LPL/WM, SLL, or MZL), received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg: Participants with CLL, who were prior BCR inhibitor naive, received new formulation of entospletinib 100 mg (1 × 100 mg tablet) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg: Participants with CLL, who were prior BCR inhibitor naive, received new formulation of entospletinib (SDD) 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD: Participants with CLL and simple progression (non-Richters), who were exposed to BTK inhibitor, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD: Participants with CLL and simple progression (non-Richters), who were exposed to PI3K inhibitor, received new formulation of entospletinib 400 mg (2 × 200 mg tablets) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD | Total
Number analyzed (Participants) | 41 | 41 | 43 | 39 | 49 | 19 | 21 | 20 | 33 | 8 | 6 | 3 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (9.6) | 66 (11.7) | 67 (14.8) | 71 (11.0) | 70 (9.8) | 69 (11.1) | 72 (10.9) | 69 (9.4) | 71 (7.4) | 61 (9.7) | 70 (8.6) | 73 (12.7) | 70 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 21 | 15 | 14 | 18 | 10 | 7 | 7 | 9 | 3 | 2 | 2 | 121
  Male | 28 | 20 | 28 | 25 | 31 | 9 | 14 | 13 | 24 | 5 | 4 | 1 | 202
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of Ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 0 | 4 | 2 | 1 | 4 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 16
    Ethnicity: Not Hispanic or Latino | 39 | 37 | 41 | 36 | 44 | 18 | 19 | 18 | 30 | 7 | 6 | 3 | 298
    Ethnicity: Not Permitted | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted=local regulators did not allow collection of Race information.
  Participants
    Race: Asian | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Race: Black or African American | 3 | 1 | 3 | 0 | 2 | 1 | 2 | 3 | 3 | 0 | 1 | 0 | 19
    Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
    Race: White/Caucasian | 37 | 39 | 37 | 36 | 45 | 18 | 19 | 17 | 27 | 8 | 5 | 3 | 291
    Race: Not Permitted | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 6
    Race: Other | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 4 | 3 | 5 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 15
  United States | 41 | 41 | 39 | 36 | 44 | 19 | 20 | 20 | 31 | 8 | 6 | 3 | 308

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Rate of Participants With CLL After BCR Targeted Therapy, MCL, and DLBCL at Week 16
Description: PFS rate was assessed by Independent Review Committee (IRC) and defined per standardized criteria (2007 Cheson criteria) (for NHL) and International Workshop on Chronic Lymphocytic Leukemia (IWCLL) criteria (for CLL), as the percentage of participants not experiencing definitive progression or death. Disease progression was defined per standardized criteria as: evidence of any new disease; worsening of nodal or extra-nodal index lesions; unequivocal increase in the size of non-index lesions or non-measurable disease, size of the liver, spleen, or other organ; and a ≥ 25% increase from nadir in either monoclonal immunoglobulin M (IgM) concentration or total serum IgM quantitation. Disease progression was defined per standardized IWCLL criteria as: evidence of any new disease; worsening of index lesions, spleen or liver, or non-index disease; and decrease in platelet count or hemoglobin that is attributable to CLL. PFS rate was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: Week 16
Population: The Full Analysis Set included all enrolled participants who took at least one dose of study drug with treatment group designated according to the planned treatment. Only participants with CLL after BCR target therapy (including CLL non-Richters, and CLL Richters participants), SDD, MCL, and DLBCL were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 43 | 39 | 33 | 8 | 6 | 3
percentage of participants | 3.6 [0.3 to 15.2] | 63.9 [45 to 77.8] | 64 [43.2 to 78.9] | 100 [100 to 100] | 20 [0.8 to 58.2] | 50 [0.6 to 91]

2. Primary Outcome: PFS Rate of Participants With CLL (Including CLL, Prior BCR Inhibitor Naive Participants), FL, and Non-FL iNHL at Week 24
Description: PFS rate was assessed by IRC and defined per standardized criteria (2007 Cheson criteria) (for NHL) and IWCLL criteria (for CLL), as the percentage of participants not experiencing definitive progression or death. Disease progression was defined per standardized criteria (2007 Cheson criteria) as: evidence of any new disease; worsening of nodal or extra-nodal index lesions; unequivocal increase in the size of non-index lesions or non-measurable disease, size of the liver, spleen, or other organ; and a ≥ 25% increase from nadir in either monoclonal IgM concentration or total serum IgM quantitation. Disease progression was defined per standardized IWCLL criteria as: evidence of any new disease; worsening of index lesions, spleen or liver, or non-index disease; and decrease in platelet count or hemoglobin that is attributable to CLL. PFS rate was analyzed using KM estimates.
Time Frame: Week 24
Population: Participants in the full analysis set were analyzed. Only participants with CLL (including CLL, prior BCR inhibitor naive participants), FL, and non-FL iNHL were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CLL: Entospletinib MM/SDD: Participants with CLL received original formulation of entospletinib 800 mg (4 × 200 mg tablets) (before amendment 8) or new formulation of entospletinib 400 mg (2 × 200 mg tablets) (after amendment 8) orally twice daily. Treatment with entospletinib was continued until disease progression or unacceptable toxicity.
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg
Number analyzed (Participants) | 41 | 41 | 49 | 19 | 21 | 20
percentage of participants | 66.9 [48 to 80.2] | 51.5 [32.8 to 67.4] | 63.5 [45.3 to 77.1] | 64.2 [33.4 to 83.6] | 81.6 [51.6 to 93.9] | 84.2 [58.7 to 94.6]

3. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Description: A treatment-emergent Adverse Event (AE) was defined as an AE that occurs in the period from the first dose of study treatment to 30 days after the last dose of study treatment or leads to discontinuation of study treatment. Participants were assessed for AEs according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03.
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 78.4 months)
Population: The Safety Analysis Set included all participants who took at least one dose of study drug with treatment group designated according to the actual treatment.
Measure: Number; unit: percentage of participants
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 41 | 41 | 43 | 39 | 49 | 19 | 21 | 20 | 33 | 8 | 6 | 3
percentage of participants | 100.0 | 100.0 | 97.7 | 97.4 | 100.0 | 100.0 | 95.2 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

4. Secondary Outcome: Percentage of Participants With Hematology Postbaseline Toxicity Grade 3 or Higher
Description: Hematology toxicity at any time postbaseline was summarized according to the NCI CTCAE, version 4.03. The most severe graded abnormality was counted for each participant per test.
  ANC = absolute neutrophil count; Hb = hemoglobin; WBC = white blood cells
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 78.4 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 41 | 41 | 43 | 39 | 49 | 19 | 21 | 20 | 33 | 8 | 6 | 3
percentage of participants
  Grade 3 ANC Decrease | 14.6 | 12.2 | 2.3 | 2.6 | 6.1 | 15.8 | 9.5 | 25.0 | 12.1 | 25.0 | 33.3 | 0
  Grade 4 ANC Decrease | 22.0 | 4.9 | 4.7 | 2.6 | 16.3 | 0 | 14.3 | 15.0 | 12.1 | 25.0 | 0 | 33.3
  Grade 3 Anemia | 14.6 | 9.8 | 14.0 | 10.3 | 22.4 | 5.3 | 19.0 | 20.0 | 27.3 | 0 | 33.3 | 33.3
  Grade 4 Anemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hb Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hb Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Leukocytosis | 34.1 | 2.4 | 0 | 5.1 | 2.0 | 52.6 | 42.9 | 40.0 | 30.3 | 25.0 | 16.7 | 0
  Grade 4 Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 WBC Decrease | 2.4 | 12.2 | 0 | 0 | 22.4 | 0 | 0 | 0 | 6.1 | 0 | 0 | 0
  Grade 4 WBC Decrease | 0 | 0 | 4.7 | 2.6 | 2.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Lymphocyte Count Decrease | 0 | 17.1 | 48.8 | 15.4 | 22.4 | 0 | 0 | 0 | 6.1 | 0 | 16.7 | 0
  Grade 4 Lymphocyte Count Decrease | 2.4 | 2.4 | 9.3 | 2.6 | 6.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Lymphocyte Count Increase | 85.4 | 9.8 | 0 | 12.8 | 6.1 | 94.7 | 85.7 | 70.0 | 63.6 | 37.5 | 33.3 | 66.7
  Grade 4 Lymphocyte Count Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Neutrophils Decrease | 14.6 | 12.2 | 2.3 | 2.6 | 10.2 | 15.8 | 9.5 | 20.0 | 12.1 | 25.0 | 16.7 | 0
  Grade 4 Neutrophils Decrease | 19.5 | 0 | 2.3 | 2.6 | 12.2 | 0 | 14.3 | 20.0 | 9.1 | 12.5 | 16.7 | 33.3
  Grade 3 Platelet Count Decrease | 7.3 | 2.4 | 2.3 | 5.1 | 6.1 | 10.5 | 4.8 | 10.0 | 15.2 | 0 | 0 | 33.3
  Grade 4 Platelet Count Decrease | 7.3 | 4.9 | 0 | 7.7 | 4.1 | 0 | 4.8 | 0 | 9.1 | 0 | 16.7 | 33.3

5. Secondary Outcome: Percentage of Participants With Serum Chemistry Toxicity Postbaseline Grade 3 or Higher
Description: Serum chemistry toxicity at anytime postbaseline was summarized according to the NCI CTCAE, version 4.03. The most severe graded abnormality was counted for each participant per test. ALT = alanine aminotransferase; ALP = alkaline phosphatase; AST = aspartate aminotransferase
Time Frame: First dose date up to the last dose date plus 30 days (maximum: 78.4 months)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 41 | 41 | 43 | 39 | 49 | 19 | 21 | 20 | 33 | 8 | 6 | 3
percentage of participants
  Grade 3 ALT Increase | 7.3 | 9.8 | 9.3 | 15.4 | 8.2 | 0 | 4.8 | 5.0 | 3.0 | 0 | 0 | 0
  Grade 4 ALT Increase | 2.4 | 9.8 | 2.3 | 7.7 | 4.1 | 0 | 0 | 5.0 | 0 | 0 | 0 | 0
  Grade 3 Hypoalbuminemia | 0 | 2.4 | 0 | 2.6 | 6.1 | 0 | 0 | 5.0 | 0 | 0 | 0 | 0
  Grade 4 Hypoalbuminemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 ALP Increase | 0 | 2.4 | 0 | 0 | 2.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 ALP Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 AST Increase | 7.3 | 12.2 | 7.0 | 10.3 | 6.1 | 0 | 0 | 5.0 | 3.0 | 0 | 0 | 0
  Grade 4 AST Increase | 0 | 4.9 | 2.3 | 2.6 | 2.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Blood Bilirubin Increase | 7.3 | 4.9 | 4.7 | 0 | 12.2 | 0 | 0 | 10.0 | 3.0 | 0 | 0 | 0
  Grade 4 Blood Bilirubin Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Creatine Kinase Decrease | 0 | 0 | 0 | 0 | 2.0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Creatine Kinase Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Creatine Kinase Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Creatine Kinase Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Creatinine | 0 | 7.3 | 2.3 | 0 | 0 | 0 | 0 | 5.0 | 0 | 0 | 0 | 0
  Grade 4 Creatinine | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Creatinine Clearance Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Creatinine Clearance Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Creatinine Clearance Increase | 9.8 | 17.1 | 2.3 | 7.7 | 4.1 | 10.5 | 4.8 | 15.0 | 12.1 | 0 | 0 | 0
  Grade 4 Creatinine Clearance Increase | 0 | 2.4 | 2.3 | 2.6 | 2.0 | 5.3 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Direct Bilirubin Decrease | 0 | 2.4 | 4.7 | 2.6 | 0 | 0 | 0 | 0 | 3.0 | 0 | 0 | 0
  Grade 4 Direct Bilirubin Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Direct Bilirubin Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Direct Bilirubin Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hyperglycemia | 9.8 | 9.8 | 4.7 | 10.3 | 16.3 | 15.8 | 9.5 | 0 | 18.2 | 0 | 16.7 | 0
  Grade 4 Hyperglycemia | 0 | 2.4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypercalcemia | 0 | 2.4 | 0 | 0 | 0 | 0 | 0 | 15.0 | 0 | 0 | 0 | 0
  Grade 4 Hypercalcemia | 0 | 2.4 | 2.3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypocalcemia | 0 | 0 | 0 | 0 | 0 | 0 | 4.8 | 0 | 3.0 | 0 | 0 | 0
  Grade 4 Hypocalcemia | 0 | 0 | 0 | 0 | 0 | 5.3 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Indirect Bilirubin Decrease | 4.9 | 2.4 | 0 | 0 | 4.1 | 0 | 0 | 10.0 | 3.0 | 0 | 0 | 0
  Grade 4 Indirect Bilirubin Decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Indirect Bilirubin Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Indirect Bilirubin Increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypermagnesemia | 2.4 | 2.4 | 2.3 | 2.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypomagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hypomagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypophosphatemia | 14.6 | 4.9 | 0 | 7.7 | 4.1 | 21.1 | 14.3 | 15.0 | 15.2 | 12.5 | 50.0 | 0
  Grade 4 Hypophosphatemia | 2.4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hyperkalemia | 4.9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hyperkalemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypokalemia | 7.3 | 9.8 | 4.7 | 0 | 2.0 | 5.3 | 4.8 | 10.0 | 3.0 | 0 | 16.7 | 0
  Grade 4 Hypokalemia | 2.4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Hyponatremia | 12.2 | 2.4 | 11.6 | 10.3 | 12.2 | 0 | 4.8 | 15.0 | 6.1 | 0 | 16.7 | 33.3
  Grade 4 Hyponatremia | 0 | 0 | 0 | 2.6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Objective Response Rate (ORR), as Assessed by IRC Per Standardized Criteria (2007 Cheson Criteria) (for NHL) and IWCLL Criteria (for CLL)
Description: ORR: percentage of participants with complete response (CR) or partial response (PR) (or very good PR [VGPR] or minor response [MR] for participants with LPL/WM). Per 2007 Cheson criteria, CR: complete resolution of all disease-related radiological abnormalities; PR: ≥50% reduction in sum of products (SPD) of the longest diameters of all index lesions, no new lesions; VGPR: >90% decrease from baseline (DFB) in IgM, and other criteria for CR met; MR: ≥25% but <50% DFB in IgM, no increase from baseline (IFB) in SPD of lesions, no new lesions. Per IWCLL, CR: lymphocytes (Ly) <4*10^9/L, no lymphadenopathy, normal spleen and liver size, absence of disease, absolute neutrophil count (ANC) >1.5*10^9/L, platelets ≥100*10^9/L, hemoglobin (Hb) >110 g/L, bone marrow at least normocellular for age; PR: ≥2 of these: ≥50% decrease in Ly, lymphadenopathy, size of liver and spleen, bone marrow infiltrates; and ≥1 of these: ANC >1500/μL, platelets ≥100,000/µL, Hb >11 g/dL.
Time Frame: From first dose date until first occurrence of CR or PR (or VGPR or MR for participants with LPL/WM) (up to approximately 7 years)
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 41 | 41 | 43 | 39 | 49 | 19 | 21 | 20 | 33 | 8 | 6 | 3
percentage of participants | 53.7 [37.4 to 69.3] | 17.1 [7.2 to 32.1] | 0 [0.0 to 8.2] | 17.9 [7.5 to 33.5] | 36.7 [23.4 to 51.7] | 26.3 [9.1 to 51.2] | 38.1 [18.1 to 61.6] | 60.0 [36.1 to 80.9] | 24.2 [11.1 to 42.3] | 75.0 [34.9 to 96.8] | 33.3 [4.3 to 77.7] | 0 [0.0 to 70.8]

7. Secondary Outcome: Duration of Response (DOR), as Assessed by IRC Per Standardized Criteria (2007 Cheson Criteria) (for NHL) and IWCLL Criteria (for CLL)
Description: DOR was defined as the interval from first documentation of CR or PR (or VGPR or MR for participants with LPL/WM) to earlier of first documentation of definitive disease progression or death from any cause. Per 2007 Cheson criteria, CR: complete resolution of all disease-related radiological abnormalities; PR: ≥50% reduction in SPD of longest diameters of all index lesions, no new lesions; VGPR: >90% DFB in IgM, and other criteria for CR met; MR: ≥25% but <50% DFB in IgM, no IFB in SPD of lesions, no new lesions. Per IWCLL criteria, CR: Ly <4*10^9/L, no lymphadenopathy, normal spleen and liver size, absence of disease, ANC >1.5*10^9/L, platelets ≥100*10^9/L, Hb >110 g/L, bone marrow at least normocellular for age; PR: ≥2 of these: ≥50% decrease in Ly, lymphadenopathy, size of liver and spleen, bone marrow infiltrates; and ≥1 of these: ANC>1500/μL, platelets ≥100,000/µL, Hb >11 g/dL. Disease progression: as defined in Outcome measure 1. DOR was analyzed using KM estimates.
Time Frame: From the date of first documentation of CR or PR (or VGPR or MR for participants with LPL/WM) to disease progression or death from any cause (up to approximately 7 years)
Population: Participants in the Full Analysis Set with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 22 | 7 | 0 | 7 | 18 | 5 | 8 | 12 | 8 | 6 | 2 | 0
months | 22 [12.7 to 36.7] | 7.6 [2.2 to NA] — Due to less number of participants with an event, upper limit of 95% CI could not be estimable. |  | 7.5 [1.9 to 14.3] | 19 [9 to 56] | 26.9 [1.7 to 42.3] | 14.9 [1.2 to 41.3] | 17. [9 to 39.2] | 8.1 [1.2 to NA] — Due to less number of participants with an event, upper limit of 95% CI could not be estimable. | 11.3 [3.4 to NA] — Due to less number of participants with an event, upper limit of 95% CI could not be estimable. | 2.7 [1.6 to 3.8] |

8. Secondary Outcome: Time to Response (TTR), as Assessed by IRC Per Standardized Criteria (2007 Cheson Criteria) (for NHL) and IWCLL Criteria (for CLL)
Description: TTR was defined as the interval from the first dose of study drug to the first documentation of CR or PR (or VGPR or MR for participants with LPL/WM). Per 2007 Cheson criteria, CR: complete resolution of all disease-related radiological abnormalities; PR: ≥ 50% reduction in SPD of the longest diameters of all index lesions, no new lesions; VGPR: >90% DFB in IgM, and other criteria for CR met; MR: ≥25% but <50% DFB in IgM, no IFB in SPD of lesions, no new lesions. Per IWCLL criteria, CR: Ly <4*10^9/L, no lymphadenopathy, normal spleen and liver size, absence of disease, ANC >1.5*10^9/L, platelets ≥100*10^9/L, Hb >110 g/L, bone marrow at least normocellular for age; PR: ≥2 of these: ≥50% decrease in Ly, lymphadenopathy, size of liver and spleen, bone marrow infiltrates; and ≥1 of these: ANC >1500/μL, platelets ≥100,000/µL, Hb >11 g/dL.
Time Frame: From the first dose of study drug to the first documentation of CR or PR (or VGPR or MR for participants with LPL/WM) (up to approximately 7 years)
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
Number analyzed (Participants) | 22 | 7 | 0 | 7 | 18 | 5 | 8 | 12 | 8 | 6 | 2 | 0
months | 3.2 (2.15) | 7.5 (4.40) |  | 4.6 (4.65) | 2.8 (2.31) | 6.4 (5.93) | 3.5 (2.39) | 6.8 (4.33) | 4.0 (2.75) | 3.4 (1.82) | 1.8 (0.05) |

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to the last dose date plus 30 days (maximum: 78.4 months); All-Cause Mortality: From enrollment up to approximately 7 years
Description: The Safety Analysis Set included all participants who took at least one dose of study drug with treatment group designated according to the actual treatment.
Arm/Group | CLL: Entospletinib MM/SDD | FL: Entospletinib MM/SDD | DLBCL: Entospletinib MM/SDD | MCL: Entospletinib MM/SDD | Non-FL iNHL: Entospletinib MM/SDD | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD
All-Cause Mortality (participants affected / at risk) | 4/41 | 3/41 | 13/43 | 6/39 | 5/49 | 0/19 | 1/21 | 1/20 | 3/33 | 1/8 | 3/6 | 1/3
Serious Adverse Events (participants affected / at risk) | 17/41 | 9/41 | 16/43 | 16/39 | 22/49 | 8/19 | 10/21 | 8/20 | 15/33 | 3/8 | 4/6 | 2/3
Other Adverse Events (participants affected / at risk) | 40/41 | 39/41 | 42/43 | 38/39 | 49/49 | 19/19 | 19/21 | 20/20 | 33/33 | 8/8 | 5/6 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CLL: Entospletinib MM/SDD (N=41) | FL: Entospletinib MM/SDD (N=41) | DLBCL: Entospletinib MM/SDD (N=43) | MCL: Entospletinib MM/SDD (N=39) | Non-FL iNHL: Entospletinib MM/SDD (N=49) | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg (N=19) | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg (N=21) | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg (N=20) | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD (N=33) | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD (N=8) | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD (N=6) | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bandaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gait inability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
H1n1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 3 | 1 | 3 | 4 | 2 | 0 | 3 | 0 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rotavirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CLL: Entospletinib MM/SDD (N=41) | FL: Entospletinib MM/SDD (N=41) | DLBCL: Entospletinib MM/SDD (N=43) | MCL: Entospletinib MM/SDD (N=39) | Non-FL iNHL: Entospletinib MM/SDD (N=49) | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 100 mg (N=19) | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 200 mg (N=21) | CLL, Prior BCR Inhibitor Naive: Entospletinib SDD 400 mg (N=20) | CLL (Non-Richters) Prior BTK Inhibitor: Entospletinib SDD (N=33) | CLL (Non-Richters) Prior PI3K Inhibitor: Entospletinib SDD (N=8) | CLL (Richters) Prior BTK Inhibitor: Entospletinib SDD (N=6) | CLL (Richters) Prior PI3K Inhibitor: Entospletinib SDD (N=3)
Anaemia (Blood and lymphatic system disorders) | 12 | 7 | 11 | 6 | 9 | 6 | 7 | 3 | 13 | 1 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglobulinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 4 | 3 | 1 | 12 | 2 | 2 | 3 | 5 | 3 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 6 | 3 | 4 | 9 | 2 | 4 | 0 | 4 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 1 | 4 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 4 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 2 | 3 | 4 | 1 | 1 | 2 | 2 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 7 | 6 | 5 | 2 | 2 | 3 | 2 | 1 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0 | 3 | 3 | 0 | 2 | 1 | 3 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 10 | 8 | 12 | 11 | 17 | 6 | 5 | 4 | 8 | 2 | 1 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 16 | 11 | 23 | 18 | 9 | 11 | 6 | 17 | 7 | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 6 | 1 | 7 | 10 | 1 | 1 | 3 | 2 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1 | 3 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 5 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 5 | 3 | 2 | 5 | 1 | 2 | 1 | 2 | 1 | 0 | 0
Gingival discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 19 | 21 | 18 | 17 | 28 | 9 | 7 | 9 | 12 | 4 | 1 | 1
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Palatal oedema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 4 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 10 | 6 | 6 | 13 | 3 | 6 | 4 | 6 | 0 | 0 | 0
Asthenia (General disorders) | 6 | 3 | 3 | 3 | 3 | 0 | 2 | 2 | 3 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 2 | 3 | 2 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chills (General disorders) | 6 | 7 | 2 | 4 | 8 | 4 | 3 | 1 | 3 | 1 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 26 | 22 | 18 | 23 | 33 | 9 | 11 | 14 | 19 | 4 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 4 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 2 | 1 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 10 | 3 | 9 | 5 | 8 | 3 | 5 | 3 | 5 | 1 | 0 | 0
Pain (General disorders) | 0 | 3 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Peripheral swelling (General disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 12 | 9 | 4 | 8 | 12 | 5 | 3 | 3 | 6 | 1 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 2 | 2 | 4 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 3 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 5 | 2 | 0 | 1 | 3 | 1 | 3 | 2 | 2 | 0 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 1 | 1 | 1 | 2 | 3 | 0 | 1 | 3 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 4 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 2 | 1 | 1 | 7 | 1 | 4 | 3 | 4 | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 7 | 3 | 2 | 3 | 5 | 2 | 1 | 3 | 3 | 1 | 0 | 0
Skin infection (Infections and infestations) | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 7 | 1 | 6 | 9 | 7 | 3 | 7 | 7 | 3 | 0 | 1
Urinary tract infection (Infections and infestations) | 8 | 5 | 5 | 4 | 3 | 5 | 3 | 3 | 4 | 0 | 2 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 4 | 5 | 0 | 2 | 2 | 2 | 2 | 0 | 3 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 6 | 0 | 2 | 3 | 6 | 1 | 1 | 2 | 3 | 1 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 2 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 7 | 4 | 7 | 5 | 0 | 2 | 2 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 7 | 6 | 5 | 2 | 0 | 2 | 2 | 1 | 2 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 5 | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 3 | 9 | 5 | 2 | 7 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 5 | 4 | 4 | 3 | 2 | 2 | 3 | 4 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
High density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 3 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Protein total decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 5 | 4 | 4 | 5 | 2 | 1 | 0 | 6 | 4 | 0 | 1 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 9 | 16 | 13 | 11 | 2 | 4 | 5 | 6 | 2 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 4 | 8 | 4 | 9 | 4 | 4 | 2 | 3 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 1 | 2 | 0 | 3 | 3 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 4 | 0 | 2 | 2 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3 | 5 | 1 | 4 | 3 | 2 | 2 | 3 | 1 | 2 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 2 | 4 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 0 | 5 | 3 | 6 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6 | 1 | 1 | 6 | 3 | 3 | 2 | 2 | 3 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 5 | 4 | 8 | 4 | 2 | 4 | 2 | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 3 | 6 | 1 | 4 | 3 | 2 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0 | 4 | 3 | 2 | 3 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 1 | 1 | 1 | 2 | 2 | 2 | 2 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 3 | 2 | 3 | 1 | 2 | 2 | 2 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 13 | 9 | 6 | 8 | 9 | 3 | 2 | 9 | 7 | 4 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 14 | 9 | 4 | 6 | 10 | 2 | 6 | 3 | 3 | 4 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 2 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 2 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 2 | 2 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 2 | 3 | 4 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 3 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 4 | 3 | 6 | 3 | 4 | 1 | 3 | 0 | 3 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 2 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 3 | 2 | 5 | 4 | 0 | 0 | 3 | 2 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 4 | 9 | 3 | 12 | 1 | 2 | 4 | 4 | 2 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 2 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 3 | 0 | 2 | 4 | 1 | 0 | 0 | 3 | 0 | 1 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Urine abnormality (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8 | 9 | 10 | 17 | 5 | 9 | 10 | 12 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 12 | 6 | 7 | 2 | 4 | 2 | 4 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 4 | 5 | 0 | 1 | 1 | 3 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 2 | 3 | 1 | 1 | 2 | 2 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0 | 4 | 6 | 1 | 2 | 0 | 2 | 2 | 0 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 2 | 5 | 2 | 2 | 3 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 4 | 1 | 4 | 6 | 0 | 4 | 1 | 3 | 1 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7 | 4 | 2 | 7 | 2 | 2 | 2 | 3 | 1 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 7 | 2 | 2 | 11 | 2 | 2 | 3 | 2 | 2 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 1 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 4 | 1 | 1 | 1 | 2 | 1 | 0 | 0
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 3 | 2 | 3 | 3 | 5 | 1 | 1 | 0 | 5 | 0 | 2 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Study was terminated prematurely due to sponsor's decision to discontinue development of entospletinib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-03-31): https://cdn.clinicaltrials.gov/large-docs/89/NCT01799889/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT01799889/SAP_001.pdf